CLINICAL TRIAL: NCT04021654
Title: What is the Future of Vulnerable New-borns
Acronym: DNNV
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0318
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-02

CONDITIONS: Preterm Birth
Keywords: Preterm birth; growth; neonatology; Pregnancy; Delivery
MeSH Terms: conditions — Premature Birth | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Data collection — Data collection of growth, neuromotor, sensorial, behavioral, and cognitive development.

SUMMARY:
The aim of this data base is to know exactly the future of a "vulnerable newborns" cared in Pontoise Hospital (In the neonatology service) and compare the information with the national data of preterm birth.

DETAILED DESCRIPTION:
The aim of this data base is to know exactly the future of a "vulnerable newborns" cared in Pontoise Hospital (In the neonatology service), it means, newborns who are in these following risk categories:

* Birth before 33 weeks of amenorrhea
* Birth between 33 and 36 weeks of amenorrhea and fetal growth retardation lower to the 3rd for the gestation age
* Perinatal anoxic-ischemia
* Other children whose birth, perinatal history or the existence of a pathology classified them in a category at risk of developmental psychomotor disorders, the co-twin of a child of the preceding groups.
* A regular follow-up is made in Pontoise hospital till the age of 7 to 8 year sold. It tries to screen growth anomalies (neuromotor, sensorial, behavioral, and cognitive or growth development) or health status. The data collect allow us to monitor these parameters and do a statistical study with them.

These information may be used to inform the parents about the future of the premature children cared at Pontoise. They also may be used to compare these children's future with the national data (EPIPAGE 2)

ELIGIBILITY:
Inclusion Criteria:

* Birth before 33 weeks of amenorrhea
* Birth between 33 and 36 weeks of amenorrhea and fetal growth retardation lower to the 3rd percentile for the gestational age.
* Perinatal anoxic-ischemia

Other children whose birth, perinatal history or the existence of a pathology classifies them in a category at risk of developmental psychomotor disorders, the co-twin of a child of the preceding groups.

Exclusion Criteria:

* Children born in normal conditions.

Ages: 1 Hour to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm bith children
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The pregnancy issues rate | 2 years
  Measure the rate of issues that occur during the pregnancy.
Delivrey issues rate | 2 years
  Measurement of the rate of issues that occur during the delivery.
% of preterm children with a failure to thrive. | 2 years
  Measurement of the % of children with a failure to thrive.

SECONDARY OUTCOMES:
Number of diseases in the children family health history. | 2 years
  Census of all diseases that may be in the children family health history

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Miler, Principal Investigator — Hôpital NOVO
Locations (1):
- Centre Hospitalier René Dubos, Pontoise, France

IPD SHARING:
Plan to Share IPD: No